CLINICAL TRIAL: NCT07107737
Title: The Role of Direct Physician Engagement in EMS Transport Refusal Rates: A Prospective Study
Brief Title: Physician Engagement in EMS Transport Refusal Rates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00134848
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-07

CONDITIONS: Refusal of Transport
Keywords: EMS transport; emergency treatment; EMS protocol
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician Consultation (Experimental): Mecklenburg EMS agency (MEDIC) crew chiefs (EMTs and/or paramedics) may decide, based on patient circumstances, to consult OMC for patients wishing to refuse care.
  Interventions: Behavioral: Physician Consultation
- Standard of Care (Active Comparator): Refusal-of-care consultation not provided to patient
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Physician Consultation — Every other month will be randomized to either Physician Consultation or Standard of Care. During the months designated for Physician Consultation, direct communication between the patient and a designated physician by phone will be implemented when a patient refuses transport in cases where the EMS clinician feels that physician consultation is warranted for further guidance. The physician will attempt to address patient concerns and provide additional medical advice.
  Arms: Physician Consultation
Behavioral: Standard of Care — Every other month will be randomized to either Physician Consultation or Standard of Care. During the months designated for Standard of Care, physician intervention will not be provided. For safety reasons, if physicians or EMS MEDIC clinicians feel that speaking with the patient is important to provide additional clinical benefit, they may do so without hesitation and can override the designated intervention month.
  Arms: Standard of Care

SUMMARY:
The primary goal of this study is to find out if patients who speak with an EMS physician over the phone are less likely to refuse care compare to patients who do not speak with an EMS physician.

DETAILED DESCRIPTION:
This study aims to assess the impact of direct physician communication on patients' decisions to refuse EMS transport. The research approach is designed to measure the influence of physician interaction on patient transport decisions in a prospective model. By conducting this research, the study team hopes to provide evidence-based recommendations for EMS protocols regarding patient engagement and refusal management.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients ≥18 years old in care of Mecklenburg EMS (MEDIC) on an emergency basis (911 call) who wish to refuse transportation to the hospital in whom MEDIC has, via existing processes and decision-making, engaged online medical control EMS Physicians for further guidance

Exclusion Criteria:

* Patients <18 years old.
* Patient refuses to speak with online medical control EMS Physicians. MEDIC or patient requests to have primary care physician.
* Lack of clinical capacity.
* Incarcerated population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Transported | Day 1
  Number of patients who agreed to be transported by EMS

SECONDARY OUTCOMES:
Number of Patients Admitted to Hospital | Day 1
  Number of patients admitted to hospital after being transported by EMS
Number of Patients Discharged from Emergency Department | Day 1
  Number of patients discharged from Emergency Department after being transported by EMS
Duration of EMS Interaction | Day 1
  Length of time from EMS arrival to the end of the patient interaction in minutes and seconds
Number of EMS Same-Day Return | Hour 24 Post Initial Call
  Number of times EMS is called again to attend to a patient who earlier refused transport

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Tyler Constantine, MD, Principal Investigator — Atrium Health Carolinas Medical Center
Locations (1):
- Atrium Health Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No